CLINICAL TRIAL: NCT02968615
Title: Simple Changes Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Yunsheng Ma, Associate professor, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00007555
Record Dates: First submitted 2016-11-07; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Overweight
Keywords: fiber; lean protein; loss weight
MeSH Terms: conditions — Overweight; Weight Loss | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fiber & protein (Experimental): A single dietary change condition that focuses exclusively on increasing fiber and protein.
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention — Participants were instructed to increase both their dietary fiber intake to 35 g/day and protein intake to 0.8 g per kilogram/day of their ideal body weight. Patients in both conditions will receive intensive dietary instruction for 6 weeks, followed by a 6 weeks maintenance phase. Participants received dietary instructions via individual and group sessions led by registered dietitians.

SUMMARY:
The investigators examined feasibility and acceptability of a non-restrictive diet focused on increasing dietary fiber and lean protein for weight loss. Fifteen obese adults enrolled in a 12-week assessment which included 6 bi-weekly individual dietary counseling sessions to attain a daily goal of higher fiber (>35 g/day) and lean protein (0.8 g per kilogram/day of individual's ideal body weight).

DETAILED DESCRIPTION:
Participants were instructed to increase both their dietary fiber intake to 35 g/day and protein intake to 0.8 g per kilogram/day of their ideal body weight. Loss of 5% of their body weight are considered to achieve the weight-loss goal. The intervention included 6 bi-weekly, 30-minute individual dietary counseling sessions over 12-weeks. Behavioral strategies including self-monitoring, problem solving, goal setting, stimulus control, food substitution, and relapse prevention were taught to assist participants in meeting their fiber and protein goals.

ELIGIBILITY:
Inclusion Criteria:

1. interested in losing weight and have a body mass index (BMI) 30-45 kg/m2;
2. ages 21 to 70;
3. able to provide informed consent;
4. physician's approval of his/her patients to participate;
5. non-smoker (given nicotine's effect on weight suppression, on HDL, and smoking cessation's effect on weight

Exclusion Criteria:

1. clinically diagnosed diabetes, or an HbA1c ≥ 6.5%;
2. an acute coronary event within the previous 6 months;
3. pregnant or lactating;
4. plans to move out of the area within the 12-week study period;
5. diagnosis of a medical condition that precludes adherence to study dietary recommendations (e.g., inflammatory bowel disease, active diverticulitis, renal disease);
6. following a low-carbohydrate, high-fat dietary regimen such as the Atkins' Diet or participating in a weight loss program;
7. previously had bariatric surgery;
8. currently using weight loss medication;
9. diagnosis of an eating disorder (anorexia nervosa, bulimia nervosa or binge eating);
10. unable to provide consent.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 weeks
  kg

SECONDARY OUTCOMES:
Total energy | 12 weeks
  kcal/day
Fiber | 12 weeks
  g/day
Protein | 12 weeks
  g/day
Saturated fat | 12 weeks
  percent of calories

CONTACTS AND LOCATIONS:
Overall Officials: Yunsheng Ma, MD, Ph.D., Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Please contact with PI